CLINICAL TRIAL: NCT06469502
Title: Comparison of the Effectiveness of Stretching and Strengthening Exercises on Pain, Functional Status, Range of Motion and Psychosocial Factors in Patients With Frozen Shoulder
Brief Title: Comparison of the Effectiveness of Stretching and Strengthening Exercises in Patients With Frozen Shoulder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Derya Celik, Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DR2024
Record Dates: First submitted 2024-06-07; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Frozen Shoulder
Keywords: frozen shoulder; exercise; stretching; strengthening
MeSH Terms: conditions — Bursitis; Motor Activity | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1-Stretching Group (Experimental): Exercise program consisting of supervised stretching exercises
  Interventions: Procedure: Stretching Exercises
- Group 2-Strengthening Group (Experimental): Exercise program consisting of supervised strengthening exercises
  Interventions: Procedure: Strengthening Exercises

INTERVENTIONS:
Procedure: Stretching Exercises — Group 1 will be included in the program consisting of stretching exercises only. Patients will receive a 6-week rehabilitation program consisting of 18 sessions of stretching exercises (3 times a week) under the supervision of a physiotherapist.
  Arms: Group 1-Stretching Group
Procedure: Strengthening Exercises — Group 2 will be included in the program consisting of strengthening exercises only. Patients will receive a 6-week rehabilitation program consisting of 18 sessions of strengthening exercises (3 times a week) under the supervision of a physiotherapist.
  Arms: Group 2-Strengthening Group

SUMMARY:
The aim of the study is to compare the effectiveness of stretching and strengthening exercises on pain, functional status, range of motion and psychosocial factors in patients with frozen shoulder.

DETAILED DESCRIPTION:
Frozen shoulder is a common disorder characterized by spontaneous shoulder pain, progressive inflammation and fibrosis of the joint capsule and loss of both active and passive glenohumeral range of motion.Exercise reduces pain, increases range of motion and function in patients with frozen shoulder. When investigators examine the literature, stretching and strengthening exercises are frequently encountered in the content of multimodal exercise programs applied clinically and at home in frozen shoulder. However, they have not been compared in isolation. Stretching is known to increase flexibility, while strengthening is often used to increase strength capacity and hypertrophy.Both exercise methods produce mechanical tension, known as a factor that stimulates anabolic metabolism and increases protein synthesis.Therefore, the aim of the study is to compare the effectiveness of stretching and strengthening exercises on pain, functional status, range of motion and psychosocial factors in patients with frozen shoulder.According to the power analysis result, 56 patients will be randomized into two groups (Group 1 =28, Group 2=28). The treatment will last for a total of 6 weeks and the follow-up period will be 6 weeks. Group 1 will be included in the program consisting of stretching exercises only. Patients will receive a 6-week rehabilitation program consisting of 18 sessions of stretching exercises (3 times a week) under the supervision of a physiotherapist. Group 2 will be included in the program consisting of strengthening exercises only. Patients will receive a 6-week rehabilitation program consisting of 18 sessions of strengthening exercises (3 times per week) under the supervision of a physiotherapist. The primary outcomes are the Quick Disabilities of the Arm, Shoulder and Hand Questionnaire (Quick DASH) and the Numeric Pain Rating Scale (NPRS), while the secondary outcomes are the American Shoulder and Elbow Surgeons Standardized Shoulder Evaluation (ASES), Shoulder range of motion, Brief Pain Inventory-Short Form (BFI-SF) and Pain Catastrophizing Scale (PCS).

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 40-65
* Clinical and radiologic diagnosis of unilateral primary frozen shoulder
* Being in frozen shoulder stages 2 and 3
* Having an ROM of less than 50% in one or more directions of shoulder flexion, abduction, external rotation compared to the unaffected shoulder
* Giving informed consent and volunteering
* To have the ability to understand evaluation scales

Exclusion Criteria:

* Neurological, cardiovascular, cerebrovascular disease
* Those with severe mental illness or impaired consciousness
* Upper extremity fractures and tumors
* Rheumatic disease
* Pathologies of cervical origin
* Untreated shoulder trauma
* Severe osteoporosis
* Previous treatment for the current complaint (physiotherapy and rehabilitation, intra-articular injection, surgery)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Quick DASH | baseline, after 6 weeks and 6 weeks follow up
  Quick Disabilities of the Arm, Shoulder, and Hand: The Quick DASH is a 11-item questionnaire used to assess upper limb functionality. The score ranges from 0 (no disability) to 100 (most severe disability).
NPRS | baseline, after 6 weeks and 6 weeks follow up
  Numeric Pain Rating Scale: The pain was measured using a NPRS. Patients are asked to rate their pain ranging from 0 to 10 (0: no pain, 10: the worst pain imaginable)

SECONDARY OUTCOMES:
ASES | baseline, after 6 weeks and 6 weeks follow up
  The American Shoulder and Elbow Surgeons Standardized Shoulder Assessment: The ASES score ranges from 0-100. Higher scores indicate better functional ability
Shoulder Range of Motion (ROM) | baseline, after 6 weeks and 6 weeks follow up
  Shoulder ROM measurements of forward flexion, abduction, and scapular plane external -internal rotation were taken using a standard goniometer. Pain-free active ROM and passive ROM were assesment.
BPI-SF | baseline, after 6 weeks and 6 weeks follow up
  Brief Pain Inventory-Short Form: The BPI is a two-factor instrument that measures pain severity and pain interference. The pain severity factor has four items, all rated on a 0-to-10 Likert scale: 0 corresponds to "no pain" and 10 corresponds to "pain as bad as you can imagine". The pain interference factor has seven items, all rated on a 0-to-10 Likert scale: 0 corresponds to "does not interfere" and 10 corresponds to "interferes completely".
PCS | baseline, after 6 weeks and 6 weeks follow up
  Pain Catastrophizing Scale: Each item is scored from 0 (never) to 4 (always), giving a total score ranging from 0 to 52. Higher scores indicate higher levels of pain catastrophizing.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes